CLINICAL TRIAL: NCT07343986
Title: Phase I Clinical Trial of Anti-CD3 × Anti-EGFR Bispecific-armed T Cells (EGFR BATs) and Low-Intensity Focused Ultrasound (LIFU) Blood-brain Barrier Opening in Patients With MGMT Unmethylated Glioblastoma (GBM)
Brief Title: Study of Low-Intensity Focused Ultrasound in Combination With Immunotherapy in Newly Diagnosed Unmethylated Glioblastoma
Acronym: BATs FUS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Focused Ultrasound Foundation (Other); NaviFUS Corporation (Industry)
Responsible Party: Principal Investigator, Camilo E. Fadul, MD, Joan and Ronald Butcher, Professor of Neurology, University of Virginia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HSR231550
Record Dates: First submitted 2025-11-25; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma (GBM)
Keywords: Focused Ultrasound; Unmethylated; Immune Therapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Arm A (Active Comparator): Arm A will have Low-Intensity Focused Ultrasound (LIFU) after infusions 4 and 8.
  Interventions: Drug: anti-EGFR bispecific-armed T cells; Device: Low-Intensity Focused Ultrasound
- Arm B (Active Comparator): Arm B will have Low-Intensity Focused Ultrasound (LIFU) after infusions 1, 4 and 8.
  Interventions: Drug: anti-EGFR bispecific-armed T cells; Device: Low-Intensity Focused Ultrasound

INTERVENTIONS:
Drug: anti-EGFR bispecific-armed T cells — IN PROGRESS
  Other Names: EGFR BATs
Device: Low-Intensity Focused Ultrasound — Low-Intensity Focused Ultrasound will be used to open the blood-brain barrier
  Other Names: LIFU

SUMMARY:
This is a phase 1 study for patients with newly diagnosed MGMT unmethylated IDH wild-type glioblastoma utilizing autologous activated T-cells armed with bispecific antibody (EGFR-BATs) that recognize the tumor. The investigators hypothesized that the combination of infusions of EGFR BATs and low-intensity focused ultrasound would induce blood-brain barrier opening and increase the permeability of the adoptive immunotherapy. The investigators will radiolabel the EGFR BATs with 89Zr-oxine for subsequent PET imaging to determine the trafficking and uptake of this approach. There is a concern that several infusions of EGFR BATs before BBB opening could change the immune tumor microenvironment that would not allow a permissive BBB after LIFU. Therefore, Arm A will have two LIFU with BBB opening after the 4th and the 8th infusion, and Arm B will have three LIFU with BBB opening after the 1st, 4th, and 8th infusions. This study will determine the safety and feasibility of the combination of low-intensity focused ultrasound (LIFU) with microbubbles BBB opening and EGFR BATs and the access of the adoptive cell immunotherapy to the tumor microenvironment to inform future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed supratentorial glioblastoma or gliosarcoma IDH wildtype and MGMT unmethylated that express EGFR (score ≥ 1 by IHC)) and confirmed by UVA pathology review.
2. Age ≥ 18 and ≤ 70 years at the time of signing informed consent.
3. Karnofsky Performance Status (KPS) ≥ 70.
4. Be willing and able to provide written informed consent for the trial.
5. Females of childbearing potential, and males, must be willing to use an effective method of contraception.
6. Maximal surgical debulking of the tumor was performed where residual contrast enhancement is 2 cm3 or less on immediate post-operative MRI. Intraoperative post-resection MRI is acceptable.
7. Able to communicate during the LIFU BBB opening procedure.
8. BBB opening target(s) must lie in non-eloquent area(s).
9. The brain tumor to be treated must be in the treatment envelope of the NaviFUS system with a minimum distance of 30 mm from the inner skull table.
10. Females of childbearing potential should have a negative serum pregnancy test. Males who are partners of females of childbearing potential must agree to use an acceptable method of contraception throughout the study and for 1 month following completion of the EGFR BATs infusions.
11. Demonstrate adequate organ function as defined in Table 1. All screening labs should be performed within 10 days before leukapheresis.

Exclusion Criteria:

1. Patients with a diagnosis of another malignancy within 2 years of being on-study. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or any type of in situ cancer. Patients must not be on any treatment for another malignancy.
2. Patients undergoing only biopsy (partial resection or greater is required).
3. Patients with cerebellar or brainstem tumors.
4. Patients with evidence of leptomeningeal dissemination or subependymal spread on initial MRI.
5. Patients with extracranial metastases.
6. Patients with evidence of acute intracranial hemorrhage.
7. Known hypersensitivity to cetuximab or another EGFR antibody.
8. Known sensitivity to gadolinium-based contrast agents.
9. Known sensitivity to Lumason® ultrasound contrast agent.
10. Alpha 1,3 Galactose IgE ("alpha gal") test result outside of the reference range (indicating likely hypersensitivity to cetuximab).
11. Patients with claustrophobia.
12. Clips, shunts, or other non-MRI compatible metallic implanted objects in the skull or the brain.
13. Evidence of active bleeding or bleeding diathesis.
14. Unable to discontinue use of anticoagulant therapy as per local standard.
15. Scalp atrophy or scars in the expected location of the ultrasound transducer.
16. Cardiac Status: Patients will be ineligible for treatment on this protocol if (before protocol entry):

    * There is a history of a recent (within one year) myocardial infarction or stroke.
    * There is a current or prior history of angina/coronary symptoms requiring medications and/or a history of depressed left ventricular function (LVEF < 45%).
    * Patient has a pacemaker.
17. There is clinical evidence of congestive heart failure requiring medical management.
18. Has Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of leukapheresis.
20. Has received any treatment for GBM besides surgery.
21. Females must not be pregnant or breastfeeding.
22. Ongoing immunosuppressive therapy except for corticosteroids
23. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
24. A patient may be excluded if, in the opinion of the treating investigator, the patient is not capable of being compliant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The safety of this treatment will be evaluated through the number of participants experiencing Grade ≥3 dose-limiting toxicities (DLTs). | 8 weeks
  The safety will be evaluated by determining the number of participants who experience Grade ≥3 DLTs according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 during EGFR BAT and LIFU BBB opening after RT/TMZ. The scale displays Grades 1 through 5 and refers to the severity of the AE. A higher grade (e.g., 5) represents a worse outcome.
The feasibility of this treatment will be determined by the proportion of participants achieving ≥75% of the recommended EGFR BATs dose | 8 weeks
  The feasibility of this treatment will be determined by calculating the proportion of participants achieving ≥75% (60 x 10^9 EGFR BATs) of the recommended Phase II EGFR BAT dose.
Incidence and severity of treatment-emergent adverse events (AEs) based on physical examination, vital signs, laboratory parameters, serum chemistry and hematology | 8 weeks
  Safety will be quantified using AE counts and severity grading per the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Physical examinations, vital signs, and laboratory studies will be recorded.
Brain uptake of 89Zr-oxine-labeled EGFR BATs measured by PET standardized uptake values (SUV) with and without LIFU BBB opening | 8 weeks
  Three PET imaging scans will be taken to quantify trafficking of labeled EGFR BATs into the GBM microenvironment. PET signal (SUV) will be compared across time points and between LIFU BBB-opened and non-opened regions.

SECONDARY OUTCOMES:
Change from baseline in peripheral immune response markers (CTL cytotoxicity) | 8 weeks
  Peripheral blood samples will be collected at baseline and at protocol-specified time points after treatment initiation. Immune response will be determined by CTL cytotoxicity. Changes from baseline will be summarized for each patient.
Change from baseline in peripheral immune response markers (IFN-γ ELISpot Counts) | 8 weeks
  Peripheral blood samples will be collected at baseline and at protocol-specified time points after treatment initiation. Immune responses will be determined by IFN-γ ELISpot Counts (SFU). Changes from baseline will be summarized for each patient.
Change from baseline in peripheral immune response markers (Th1/Th2 serum cytokine concentrations) | 8 weeks
  Peripheral blood samples will be collected at baseline and at protocol-specified time points after treatment initiation. Immune responses will be determined by Th1/Th2 serum cytokine concentrations. Changes from baseline will be summarized for each patient.
PET-based quantification of 89Zr-oxine-labeled EGFR BAT trafficking across the BBB and into the GBM microenvironment after infusions and Low Intensity Focused Ultrasound (LIFU). | 8 weeks
  PET imaging will be used to measure radiotracer uptake (SUV) in the brain and tumor regions following infusions of 89Zr-labeled EGFR BATs. PET SUV after the 1st infusion's LIFU will be compared to the PET SUV after the 4th and the 8th infusion's LIFU.
PET-based quantification of 89Zr-oxine-labeled EGFR BAT trafficking across the BBB and into the GBM microenvironment with versus without Low Intensity Focused Ultrasound (LIFU). | 8 weeks
  PET imaging will be used to measure radiotracer uptake (SUV) in the brain and tumor regions following infusions of 89Zr-labeled EGFR BATs. PET scans with and without LIFU BBB opening will be compared within patients and between study arms (Arm A vs Arm B). Specifically, PET SUV of patients who had LIFU after the infusion will be compared to patients who did not have LIFU after the infusion.
Quantitative levels of circulating tumor DNA (ctDNA) | 8 weeks
  Peripheral blood will be collected before the 1st, 4th, and 8th EGFR BAT infusions and 1-2 hours after LIFU BBB opening. ctDNA concentration will be measured and expressed as absolute values and change from baseline.
Quantitative levels of antibodies against tumor-associated antigens (IgG anti-EGFR and IgG anti-HER2) | 8 weeks
  Peripheral blood will be collected before the 1st, 4th, and 8th EGFR BAT infusions and 1-2 hours after LIFU BBB opening. The serum concentration of IgG anti-EGFR and IgG anti-HER2 will be measured by Enzyme-Linked Immunosorbent Assay (ELISA).
Progression-free survival (PFS) measured using modified Response Assessment in Neuro-Oncology (RANO) criteria. | From date of surgery to date of first documented progression, assessed up to 104 weeks.
  PFS will be defined as the time from surgery to the earliest date of confirmed radiographic or clinical progression determined by MRI and using modified RANO criteria. Progression will be determined by ≥25% increase in bidirectional product or ≥40% volumetric increase, development of new measurable disease, or clinical deterioration attributable to tumor. RANO scoring evaluates brain tumor response to treatment using MRI scans, categorizing the outcomes Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD) based on changes in tumor size (measured by Sum of Perpendicular Diameters or volumetric methods).
Overall survival (OS) | From date of surgery to date of documented death, assessed up to 104 weeks.
  OS will be defined as the time from surgery to death from any cause.
Correlation between immune response measures and clinical outcomes | From baseline until 1-year post-treatment completion
  Immune biomarkers (CTL cytotoxicity, IFN-γ ELISpot counts, Th1/Th2 cytokines, antibodies, ctDNA) will be correlated with clinical outcomes, including objective radiographic response (modified RANO), PFS, and OS. Associations will be evaluated using continuous and categorical analyses.
Objective response rate (ORR) per modified Response Assessment in Neuro-Oncology (RANO) criteria | From baseline until 1-year post-treatment completion
  ORR will be calculated as the proportion of participants achieving confirmed complete response or partial response, defined by modified RANO volumetric or bidimensional thresholds. RANO scoring evaluates brain tumor response to treatment using MRI scans, categorizing the outcomes Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD) based on changes in tumor size (measured by Sum of Perpendicular Diameters or volumetric methods).
Incidence and severity of adverse events (AEs) and laboratory abnormalities | From baseline through 30-days post-treatment completion
  Safety will be assessed through physical examinations, vital signs, laboratory studies, serum chemistry and hematology. AEs will be graded using CTCAE v5.0. Counts and severity grades will be summarized over the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Camilo Fadul, M.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fadul CE, Thakur A, Kim J, Kassay-McAllister J, Schalk D, Lopes MB, Donahue J, Purow B, Dillon P, Le T, Schiff D, Liu Q, Lum LG. Phase I study targeting newly diagnosed grade 4 astrocytoma with bispecific antibody armed T cells (EGFR BATs) in combination with radiation and temozolomide. J Neurooncol. 2024 Jan;166(2):321-330. doi: 10.1007/s11060-024-04564-y. Epub 2024 Jan 23. PMID 38263486